CLINICAL TRIAL: NCT02870569
Title: A Multicenter, Randomized, Open-Label,Phase 2 Trial of Donafenib in 131I-Refractory Differentiated Thyroid Cancer
Brief Title: Phase 2 Trial of Donafenib in 131I-Refractory Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG01N-1271
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2017-08

CONDITIONS: Differentiated Thyroid Cancer
MeSH Terms: interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donafenib1 (Experimental): This is the lower dose group. Donafenib 200mg bid
  Interventions: Drug: Donafenib 200mg
- Donafenib2 (Active Comparator): This is the higher dose group. Donafenib 300mg bid
  Interventions: Drug: Donafenib 300mg

INTERVENTIONS:
Drug: Donafenib 200mg — Donafenib is an oral multikinase inhibitor with antiproliferative and antiangiogenic effects.The arm is the lower dose one.
  Other Names: lower dose
  Arms: Donafenib1
Drug: Donafenib 300mg — Donafenib is an oral multikinase inhibitor with antiproliferative and antiangiogenic effects.The arm is the higher dose one.
  Other Names: higher dose
  Arms: Donafenib2

SUMMARY:
Donafenib for advanced 131I-refractory/resistant differentiated thyroid cancer(DTC).

DETAILED DESCRIPTION:
This phase 2 study of donafenib, an oral multikinase inhibitor that targets Raf kinase and receptor tyrosine kinases, is to assess efficacy and safety in patients with 131I-refractory/resistant differentiated thyroid cancer.The study is a randomised,multicentre,open-label study.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastases thyroid cancer;
* Subjects must have histologically or cytologically confirmed diagnosis of one of the following differentiated thyroid cancer (DTC) subtypes: papillary thyroid cancer (PTC),follicular thyroid cancer (FTC) or Hurthle cell ;
* Measurable disease meeting the following criteria and confirmed by central radiographic review:

  1. At least 1 lesion of greater than or equal to 1.0 cm in the longest diameter for a non-lymph node or greater than or equal to 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computerized tomography.
  2. Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radio-frequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion;
  3. Bone metastases lesion is non-measurable.
* Subjects must show evidence of disease progression within 14 months prior to signing informed consent, according to RECIST 1.1 assessed and confirmed by central radio-graphic review of CT scans.
* Subjects must be 131I-refractory / resistant as defined by at least one of the following:

  1. One or more measurable lesions that do not demonstrate iodine uptake on any radio-iodine scan
  2. One or more measurable lesions that has progressed by RECIST 1.1 within 14 months of 131I therapy, despite demonstration of radio-iodine avidity at the time of that treatment by pre-treatment scanning.
  3. Cumulative activity of 131I of >600 mCi or 22 gigabequerels (GBq), with the last dose administered at least 6 months prior to study entry
* Subjects may have not received molecular targeted therapy;
* Subjects with known brain metastases who have completed whole brain radiotherapy, stereotactic radiosurgery or complete surgical resection, will be eligible if they have remained clinically stable, asymptomatic and off of steroids for one month
* Subjects must tolerate to thyroxin ,and TSH suppression (TSH less than 0.1 mU/mL);
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~2；
* Life expectancy of at least 3 months;
* Adequate bone marrow function:

  1. Absolute neutrophil count (ANC) greater than or equal to 1500/mm3;
  2. Platelets greater than or equal to 100,000/mm3 ;
  3. Hemoglobin greater than or equal to 9.0g/dL
* Adequate blood coagulation function:

  1. Prothrombin time(PT)≤17s;
  2. Activated prothrombin time(APTT)≤47s;
  3. International Normalized Ratio(INR)≤2.
* Adequate liver function:

  1. Bilirubin less than or equal to 1.5 x the upper limit of normal(ULN) ;
  2. Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 2.5 x the upper limit of normal (ULN).
* All females must have a negative serum or urine pregnancy test. Females of childbearing potential and male subjects who are partners of women of childbearing potential must use or their partners must use a highly effective method of contraception;
* Voluntary provision of written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

* Anaplastic or Medullary carcinoma of the thyroid;
* Prior treatment to sorafenib or other molecular targeted drugs;
* Subjects who have received any chemotherapy or extra radiotherapy within 30 days prior to the first dose of study drug and should have recovered from any toxicity related to previous anti-cancer treatment;
* Major surgery within 30 days prior to the first dose of study drug;
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina; myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment;
* Active infection (any infection requiring treatment);
* Active malignancy (except for differentiated thyroid carcinoma, or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months;
* Known intolerance to any of the study drugs (or any of the excipients);
* All chemotherapy or radiation-related toxicities must have resolved to less than Grade 2 severity, except alopecia and infertility;
* Adequately controlled blood pressure with or without antihypertensive medications, defined as BP less than 140/90 mmHg using at least 2 kinds of medicine;
* Adequate renal function defined as calculated creatinine clearance less than or equal to 60 mL/min per the Cockcroft and Gault formula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07-02 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | From randomization of the first subject until the last subject complete 24 months treatment
  ORR is defined as the percentage of subjects with total number of Complete Response(CR)+total number of Partial Response(PR).

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization of the first subject until the last subject complete 48 months treatment
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact
Progression-free Survival (PFS) | From randomization of the first subject until the last subject complete 24 months treatment
  PFS was defined as the time from date of randomization to disease progression radiological or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.
Safety variables will be summarized using descriptive statistics based on adverse events collection | From randomization of the first subject until the last subject complete 24 months treatment
  Patients with adverse events/all patients *100%
Disease Control Rate(DCR) | From randomization of the first subject until the last subject complete 24 months treatment
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun D, Zhang X, Jin X, Shi C, Sun Y, Zhang Y, Liang J, Lin Y. BRAFV600E mutation is associated with better prognoses in radioactive iodine refractory thyroid cancer patients treated with multi-kinase inhibitors: a retrospective analysis of registered clinical trials. Thyroid Res. 2025 Feb 10;18(1):5. doi: 10.1186/s13044-025-00223-0. PMID 39924483
- [Derived] Lin YS, Yang H, Ding Y, Cheng YZ, Shi F, Tan J, Deng ZY, Chen ZD, Wang RF, Ji QH, Huang R, Li LF. Donafenib in Progressive Locally Advanced or Metastatic Radioactive Iodine-Refractory Differentiated Thyroid Cancer: Results of a Randomized, Multicenter Phase II Trial. Thyroid. 2021 Apr;31(4):607-615. doi: 10.1089/thy.2020.0235. Epub 2020 Oct 15. PMID 32907500